CLINICAL TRIAL: NCT06011525
Title: Prevention of Alopecia in Patients With Localised Breast Cancer by Scalp cooLing vs Cooling Mask: a Randomised Controlled Trial With Medico-economic Evaluation
Brief Title: Prevention of Alopecia in Patients With Localised Breast Cancer
Acronym: ICELAND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-A00769-36
Record Dates: First submitted 2023-08-03; First posted 2023-08-25 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy-induced Alopecia
Keywords: alopecia; chemotherapy-induced
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard cold-cap (Active Comparator): Patients will benefit from the prevention of chemo-induced alopecia using the standard cold cap device throughout the course of anthracycline- and taxane-based chemotherapy.
  This device will be supplemented by a compression bandage to add to the vasoconstriction action of the cold, the compression of the bandage on the scalp and thus optimise the effectiveness of the device.
  Interventions: Other: standard cold cap
- scalp-cooling technique (Experimental): Patients will benefit from the prevention of chemo-induced alopecia using the standard cold cap device throughout the course of anthracycline- and taxane-based chemotherapy.
  Interventions: Other: scalp-cooling technique

INTERVENTIONS:
Other: standard cold cap — Standard cold-cap applied throughout anthracycline- and taxane-based chemotherapy treatment.
  This device will be supplemented by a compressive bandage in order to add to the vasoconstriction action of the cold, the compression of the bandage on the scalp and thus optimise the efficacy of the device.
  Arms: standard cold-cap
Other: scalp-cooling technique — Scalp-cooling technique applied throughout anthracycline- and taxane-based chemotherapy treatment
  Arms: scalp-cooling technique

SUMMARY:
The prevention of chemotherapy-induced alopecia (CIA) is still imperfectly managed in France. Strengthening the evidence base on the benefits of strategies to prevent CIA, based on robust methodologies, remains a prerequisite for better integration of appropriate supportive care for patients receiving chemotherapy.

This research should provide new knowledge on the benefits of scalp refrigeration during anthracycline- and taxane-based chemotherapy in preventing ACI, for each of the 2 refrigeration techniques. In addition to effectiveness in preventing ACI, quality of life, self-image and satisfaction with care will be assessed by patients during and after chemotherapy. The medico-economic aspects will also be assessed for each of the two refrigeration modalities. The results of the various proposed assessments will be used to guide the choice between these two techniques for preventing ACI.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Female
* Histologically proven diagnosis of localised, non-metastatic breast cancer
* Indication for neo-adjuvant or adjuvant anthracycline and taxane chemotherapy (3 or 4 EC100 followed by 3 Docetaxel or 3 or 4 EC100 plus 9 to 12 Paclitaxel); HER-positive status is not a non-inclusion criterion.
* Patient willing to be photographed to assess IFA
* Fluency in French
* Patient affiliated to a social security scheme
* Signature of informed consent

Exclusion Criteria:

* History of neck pain
* Pre-existing alopecia
* Participation in another trial
* Dermatosis of the scalp
* Contraindication to scalp cooling
* History of migraines, stroke or hyperthyroidism
* History of scalp metastases
* Sensitivity to cold, cold agglutinin disease, cryoglobulinaemia, cryofibrinogenaemia or post-traumatic cold dystrophy.
* Malignant haemopathies
* History of chemotherapy treatment
* Indication for cerebral irradiation
* Pregnant or breast-feeding patient
* Raynaud's syndrome

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2026-09-03 (Estimated); Study Completion 2028-09-08 (Estimated)

PRIMARY OUTCOMES:
Compare the grade of the patient alopecia. | At 6 months after treatment start
  The grade of patient alopecia will be be evaluated by NCI-CTCAE

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - IUCT-Oncopole, Toulouse